CLINICAL TRIAL: NCT02511886
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Determine the Maximum Tolerated Dose of Arbaclofen Placarbil in Subjects With Alcohol Use Disorder
Brief Title: A Dose-Escalation Study to Determine the Maximum Tolerated Dose of Arbaclofen Placarbil in Subjects With Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RB-US-14-0001
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Alcohol Use Disorder
Keywords: Alcoholism; Alcohol Abuse; Alcohol Addiction; Alcohol Dependence; Alcohol Induced Disorders; Alcoholic Intoxication
MeSH Terms: conditions — Alcoholism; Alcohol-Induced Disorders; Alcoholic Intoxication | interventions — arbaclofen placarbil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arbaclofen Placarbil (AP) (Experimental): Orally administered Arbaclofen Placarbil (AP) sustained release (SR) tablets
  Interventions: Drug: Arbaclofen Placarbil
- Placebo (Placebo Comparator): Subjects remain on placebo for entire study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arbaclofen Placarbil — Arbaclofen Placarbil
  Arms: Arbaclofen Placarbil (AP)
Drug: Placebo — Placebo matched tablets
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This study will determine the maximum tolerated dose (MTD) of arbaclofen placarbil (AP) in the treatment of subjects with Alcohol Use Disorder (AUD). For every two subjects receiving AP, one subject will receive placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled dose-escalation study to determine the MTD of AP in subjects with AUD. Eighteen (18) subjects will be randomized to receive either AP or placebo in a 2:1 ratio; ie, 12 subjects will be assigned to AP and 6 will be assigned to placebo. Efforts will be made to enroll all subjects in the same period of time at one clinical center. The expected maximum duration of participation for each subject is 11 weeks and will consist of up to a 3-week screening period, up to a 30-day residential (inpatient) treatment period, up to a 4-week non-residential (outpatient) treatment period, and an end of study / early termination clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age.
2. Diagnosis of AUD confirmed by the Mini-International Neuropsychiatric Interview.
3. For those requiring medical detoxification from alcohol, subjects will be required to have completed a program for detoxification from alcohol within 4 days prior to screening.
4. Provide written informed consent prior to any study-specific procedures.
5. Self-report of at least 2 heavy drinking days per week in each of the 4 weeks prior to the screening interview.
6. Willing to abstain from drinking for the time he/she is participating in the study.
7. Able to identify at least 1 "locator" person to assist study staff in tracking the subject for the non-residential clinic days.
8. Able to read, speak, and understand English and be willing to cooperate with study procedures.
9. For female subjects, women of childbearing potential must have a negative pregnancy test prior to enrollment and must agree to use a medically acceptable means of contraception from screening through at least 3 months after the last dose of IMP. Male subjects with female partners of childbearing potential must agree to use medically acceptable contraception from informed consent through at least 3 months after the last dose of IMP. Male subjects must also agree not to donate sperm during the study and for 3 months after receiving the last dose of IMP (Investigational Medicinal Product).

Exclusion Criteria:

1. Has present symptoms or history of any of the following disorders:

   * Schizophrenia
   * Schizoaffective Disorder
   * Delusional Disorder
   * Bipolar I Disorder
   * Any mood disorder with psychotic features or any psychotic disorder
   * Anorexia Nervosa
   * Bulimia Nervosa
   * Post-Traumatic Stress Disorder that could interfere with the study
   * Any Personality Disorder that could interfere with the study
2. Current diagnosis of any substance use disorder, except for nicotine, cannabis (mild or moderate), or alcohol.
3. Positive result for any prohibited medication.
4. History of suicidal ideation within 30 days prior to providing written informed consent.
5. History of seizures or delirium tremens.
6. Intention to initiate or continue additional formal alcohol-related treatment, including pharmacotherapy, during the active treatment period.
7. Have had inpatient treatment for a non-alcohol substance use disorder in the 12 weeks prior to informed consent.
8. Total bilirubin >1.5× the upper limit of normal (ULN), alanine aminotransferase (ALT) >3×ULN, aspartate aminotransferase (AST) >3×ULN, serum creatinine >2×ULN, international normalized ratio (INR) >1.5×ULN, lipase >3×ULN, amylase >3×ULN, or any abnormal pancreatic enzyme value above ULN that is associated with clinically significant active pancreatic disorder.
9. Creatinine clearance of <80 mL/min, as calculated according to the Cockcroft-Gault equation.
10. Hemoglobin at screening of <11.5 g/dL (for females) or <12.5 g/dL (for males).
11. Body mass index (BMI) >30.
12. Diagnosed with unstable medical disorders that could increase the potential risk of study treatment or interfere with study participation, including the following:

    1. Abnormal cardiac conditions, including:

       * Uncontrolled hypertension.
       * History of myocardial infarction in the last year or any prior history of myocardial infarction with active complication.
       * Syncopal event within the past year.
       * Congestive heart failure.
       * Angina pectoris.
       * QTcF (QT Fridericia-corrected) ≥450 msec for males and ≥470 msec for females at screening or randomization.
       * Clinically significant abnormal finding on the physical exam or 12-lead ECG.
    2. Diabetes mellitus (type 1 or 2) fulfilling any of the following criteria:

       * Glycosylated hemoglobin (HbA1c) >7.5% at screening.
       * Uncontrolled diabetes mellitus.
13. Have any other clinically significant abnormal laboratory result
14. Must not have donated blood or have had any therapeutic phlebotomy (in an amount >300 mL) or received blood transfusion within 90 days preceding enrollment.
15. Must not have a history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system disorder (eg, Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system (CNS), or a history of significant head trauma within the past 2 years, or currently receiving anticonvulsant therapy for any reason.
16. Must not have acquired immunodeficiency syndrome (AIDS).
17. Have any other active medical condition or organ disease that may either compromise subject safety or interfere with the safety and/or outcome evaluation of the IMP.
18. History or presence of allergic or adverse response (including rash or anaphylaxis) to baclofen or any ingredient of the IMP.
19. Have used baclofen within 30 days prior to informed consent.
20. Taking medications which may be expected to significantly interfere with the metabolism or excretion of AP, may be associated with a significant drug interaction with AP, or may pose a significant risk to the subject's participation in the study.
21. Participation in an interventional clinical study within 30 days prior to informed consent.
22. Use of exclusionary drugs (e.g. antipsychotics, anticonvulsants, benzodiazepines, naltrexone, acamprosate).
23. Site staff or subjects affiliated with, or a family member of, site staff directly involved in the study.
24. Be unable to comply fully with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Arbaclofen Placarbil | Up to 30 day residential (inpatient) treatment period
  A data monitoring committee (DMC) will review and make a recommendation to stop dosing escalation based on the review of the unblinded AE and safety assessments or when at least one subject on active investigational product experiences an SAE related to the investigational product. The MTD and the dosage that will not be exceeded in the further development of this compound will be based upon a comprehensive review of the safety data.
Maximum Observed Plasma Concentration of Arbaclofen Placarbil (AP) (Cmax) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20, and 24 hours post-dose (predose day 2); and prior to dose of AP on days 6, 12, 18, and 24 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours post dose
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods
Time to Maximum Observed Plasma Concentration of Arbaclofen Placarbil (AP) (Tmax) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20, and 24 hours post-dose (predose day 2); and prior to dose of AP on days 6, 12, 18, and 24 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours post dose
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods
Area Under the Concentration -Time Curve from time 0 to the time of the last quantifiable plasma concentration (AUClast) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post dose
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods
Area Under the Concentration -Time Curve from time 0 extrapolated to infinite time (AUCinf) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post dose
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods
Area Under the Concentration -Time Curve from time 0 to 12 hours post dose(AUC0-12) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post dose
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods
Apparent Terminal Plasma Half-Life (t 1/2) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods
Apparent Terminal Phase Rate Constant | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post dose
  Apparent terminal rate constant (1/h), determined by linear regression of the terminal points of the log-linear concentration-time curve. Visual assessment will be used to identify the terminal linear phase of the concentration-time profile. A minimum of 3 data points will be used for determination.
Percentage of AUCinf obtained by extrapolation (%AUCex) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post dose
  If the extrapolated area is greater than 20% of AUCinf, then AUCinf will be listed but not included in summary presentations or statistical analyses
Apparent Oral Clearance (CL/F) | Prior to the initial dose of AP on day 1, 6, 12, 18, 24 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post dose
  Calculated as Dose/AUCinf
Apparent Volume of Distribution (Vz/F) | Prior to the initial dose of AP on day 1 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8,10, 12, 16, 20 hours post dose
  Calculated as Dose/apparent terminal phase rate constant * AUCinf
Area Under the Plasma Concentration-Time Curve From Time Zero To The End of Dosing Interval (AUCtau) | Prior to dose of AP on days 6, 12, 18, and 24 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours post dose
  Area Under the Plasma Concentration-Time Curve From Time 0 to the End of the Dosing Interval
Minimum Observed Plasma Concentration (Cmin) | Prior to dose of AP on days 6, 12, 18, and 24 and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours post dose
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods
Pre-Dose Plasma Concentration (Ctrough) | Prior to dose of AP on days 6, 12, 18, 19, 20, 21, 22, 23, and 24 hours post dose
  Blood samples will be obtained and plasma concentrations determined using a validated liquid chromatography with tandem mass spectrometry methods

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Serious or Non-Serious Adverse Events | Up to 11 weeks
  A non-serious adverse event is any untoward medical occurrence. A serious adverse event is any adverse event that meets one or more of the following: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important event, as defined in the protocol
Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 11 weeks
  All events of suicide-related behavior will be carefully monitored. These include emergence or significant worsening of reported suicidal ideation, plans, suicide attempts, and completed suicides. The C-SSRS will be used by the Investigator in the assessment of suicide risk.
The Obsessive-Compulsive Drinking Scale (OCDS) | Up to 11 weeks
  All continuous outcome measures including time to event endpoints collected will be summarized using descriptive statistics (n, mean, standard deviation (SD), median, min, and max). Categorial variables will be summarized using frequencies.
Hospital Anxiety and Depression Scale (HADS) | Up to 11 weeks
  The HADS is a 14-item scale that generates original data. Seven f the items relate to anxiety and 7 relate to depressive symptoms. Zigmond and Snaith created this outcome measure specifically to avoid reliance on aspects of these conditions that are also common somatic symptoms of illness; eg, fatigue, insomnia, or hypersomnia
Alcohol Liver Biomarkers (Carbohydrate Deficient Transferrin and Gamma Glutamyl Transferase | Up to 11 weeks
  Blood samples will be collected and sent to the central laboratory.
Timeline Follow Back (TLFB) Interview for Cigarette and Alcohol Use | Up to 11 weeks
  The TLFB interview is a method to assess recent alcohol use and will be administered by an interviewer to estimate retrospectively their alcohol use (frequency and number of drinks consumed)
Short Inventory of Problems-Revised (SIP-R) | Up to 11 weeks
  The SIP-R is a 17 item self-reported inventory of adverse consequences associated with drug and alcohol use developed by Blanchard (2003). The SIP instructs participants to indicate how often each of the listed consequences has occurred during the past month on a 4-point scale (0-3). Item responses are summed to produce a total score and 5 subscale scores

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Development Manager, Study Director — Indivior Inc.
Locations (1):
- Research Centers of America, Oakland Park, Florida, United States

IPD SHARING:
Plan to Share IPD: No